CLINICAL TRIAL: NCT04179760
Title: A Randomized, Phase I/II Trial to Evaluate the Safety and Efficacy of SCM-AGH in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Safety and Efficacy of SCM-AGH in Subjects With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCM Lifescience Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADT2002
Record Dates: First submitted 2019-11-20; First posted 2019-11-27 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Phase I: Multicenter in Korea, Randomized, Open-label, Parallel arm Phase II: Multicenter in Korea, Double-blind, Placebo-controlled, Parallel arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCM-AGH (Experimental): * Ingredient: Allogeneic human bone marrow-derived mesenchymal stem cells
  * Dose: 1x10^6 cells/Kg
  Interventions: Biological: SCM-AGH
- Placebo (Placebo Comparator): 3 times with 2-week intervals by IV infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SCM-AGH — SCM-AGH will be administrated 3 times with 2-week intervals by IV infusion to subjects at Weeks 0, 2 and 4 (Visits 2, 3 and 4).
  Arms: SCM-AGH
Other: Placebo — Placebo will be administrated 3 times with 2-week intervals by IV infusion to subjects at Weeks 0, 2 and 4 (Visits 2, 3 and 4).
  Arms: Placebo

SUMMARY:
This study consists of two phases (Phase I and Phase II). Phase II will be conducted sequentially after the safety of SCM-AGH is secured in Phase I.

Phase I: Multicenter in Korea, Randomized, Open-label, Parallel arm Phase II: Multicenter in Korea, Double-blind, Placebo-controlled, Parallel arm

DETAILED DESCRIPTION:
Phase I (Multicenter, Randomized, Open-label, Parallel arm Design) Twenty subjects with moderate to severe Atopic Dermatitis(AD) are planned to be enrolled from 6 sites in Korea and administered with SCM-AGH by intravenous (IV) infusion 3 times at two-week intervals and evaluated for safety during the safety evaluation period (12 weeks after first infusion).

Phase II (Multicenter, Double-blind, Placebo-controlled, Parallel arm) Phase II of the study is randomized, double-blind, placebo-controlled, parallel arm comparison study in adult subjects with moderate to severe AD. 72 subjects with moderate to severe AD are planned to be enrolled from 6 sites in Korea. Following up to a 4-week Screening period, subjects will be randomly assigned to one of the following treatment arms: SCM-AGH or placebo in the ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are males or females aged >= 19 years
2. Subjects who are diagnosed with Atopic Dermatitis (AD) based on the Eichenfield revised criteria of Hannifin and Rajka that

   1. has been present for at least 1 year before the Screening visit, and
   2. have chronic AD symptoms continually for at least 6 months before Screening visit
3. Subjects who have moderate to severe AD (EASI ≥16) at the Screening visit and Baseline visit
4. Subjects who have IGA score ≥3 at the Screening and Baseline visits
5. Subjects who have at least 10% of total body surface area affected by AD at the Screening and Baseline visits
6. Subjects who can give written informed consent
7. Subjects must have applied a stable dose of a bland emollient to affected areas for at least 7 days before the Baseline visit and be willing to continue for the duration of the study
8. Male subjects must abstain from heterosexual activities or agree to use a condom through 30 days after the final dose of study drug. Women of childbearing potential (WOCBP) must abstain from heterosexual activities or agree to use effective contraception through 30 days after the final dose of study drug.

Effective contraception for males and/or WOCBP includes:

* Blockage methods - spermicides and condoms/spermicides and vaginal diaphragm for contraception, vaginal sponges or cervical cap (where available)
* Oral contraceptives ("the pill") for at least 1 month
* Depot or injectable birth control or implantable contraception (e.g., Implanon)
* Intrauterine device (IUD)
* Documented evidence of surgical sterilization at least 6 months prior to Screening visit i.e., tubal ligation or hysterectomy for women or vasectomy for men
* Women who are post-menopausal, as documented by measurement of follicle stimulating hormone

Exclusion Criteria:

1. Systemic infection or local infection requiring prohibited medications at Screening visit
2. Subjects who underwent the following treatments within 4 weeks prior to Baseline visit or are scheduled to receive the following treatments within 4 weeks from Baseline at the discretion of investigator:

   1. Use of immunosuppressive/ immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ (interferon-gamma), Janus kinase inhibitors, azathioprine, methotrexate)
   2. Phototherapy for AD
   3. Any other systemic therapy used to treat AD or symptoms of AD (approved or off-label use)
3. Use of topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within at least 2 weeks prior to Baseline
4. History of anaphylaxis to any biologic therapy or vaccine
5. History of Guillain-Barré syndrome
6. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained
7. Any allergen immunotherapy within 4 months prior to or throughout the study
8. A value outside the specified range of 90 mmHg - 140 mmHg for systolic blood pressure and 50 mmHg -90 mmHg for diastolic blood pressure (both inclusive) at Screening (can be repeated once at Screening as per Principal Investigator's [PI's] discretion).
9. Receipt of live vaccines within 12 weeks prior to Baseline
10. Receipt of the following biologics:

    1. Cell depleting agents such as rituximab: within 6 months prior to Baseline or within time to return of lymphocyte count to normal, whichever is longer
    2. Other biologics: within 5 half-lives or within 16 weeks prior to Baseline, whichever is longer
11. Active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus (HCV)
12. Female subjects who are pregnant or lactating or female subjects of childbearing potential who have a pregnancy plan or do not agree to use acceptable methods of contraception, excluding females who are in post-menopausal or surgically infertile (bilateral tubal ligation, bilateral oophorectomy or complete hysterectomy)
13. Receipt of any investigational drugs within 8 weeks prior to baseline, within 5 half lives of investigational drug or participated in any clinical trials of medical device
14. Diagnosed with either primary or recurrent malignancy within 5 years from Screening
15. Liver malfunctions with aspartate aminotransferase (AST) / alanine aminotransferase (ALT) level >2x upper limit of normal (ULN) at Screening
16. Renal malfunctions with creatinine level >2x ULN at Screening
17. QTc (corrected QT interval) prolongation >470 msec or other significant ECG abnormality noted within 14 days of treatment
18. History of hypersensitivity to antibiotics and antimicrobial agents
19. History of significant Adverse Events (AEs) during stem cell therapies
20. Allergic or hypersensitivity reaction to the IP (Investigational Product), drug of similar class or ingredients [bovine serum, dimethyl sulfoxide (DMSO)]
21. Failure to comply with emollient application instructions prior to baseline, per diary
22. Subjects who, in the opinion of the investigator, have other unstable intercurrent diseases that confound safety and efficacy assessment
23. Planned or anticipated major surgical procedure during the subject's participation in this study
24. Subjects who, in the opinion of the investigator, would be non-compliant with the visit schedule of study procedures

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
over 50% reduction ratio of Eczema Area and Severity Index (EASI) as contrasted with baseline value (EASI-50) | Week 12
  An EASI score is a tool used to measure the extent (area) and severity of atopic eczema (Eczema Area and Severity Index). The minimum EASI score is 0 and the maximum EASI score is 72. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Score change from Baseline in Eczema Area and Severity Index(EASI) score | Weeks 4, 8, 12, 16, 20 and 24
  An EASI score is a tool used to measure the extent (area) and severity of atopic eczema (Eczema Area and Severity Index). The minimum EASI score is 0 and the maximum EASI score is 72. Higher scores mean worse outcome.
Percentage of subjects who have EASI-75 (improvement of ≥75% in EASI score from Baseline) | Weeks 12, 16, 20 and 24
  An EASI score is a tool used to measure the extent (area) and severity of atopic eczema (Eczema Area and Severity Index). The minimum EASI score is 0 and the maximum EASI score is 72. Higher scores mean worse outcome.
Percentage of subjects who have EASI-90 (improvement of ≥90% in EASI score from Baseline) | Weeks 12, 16, 20 and 24
  An EASI score is a tool used to measure the extent (area) and severity of atopic eczema (Eczema Area and Severity Index). The minimum EASI score is 0 and the maximum EASI score is 72. Higher scores mean worse outcome.
Percentage of subjects who have the Investigator's Global Assessment (IGA) score of 0 or 1 | Weeks 12, 16, 20 and 24
  This assessment is the overall investigator's overall global assessment for the whole body. Minimum 0 to Maximum 4. 0 means No inflammatory signs of atopic dermatitis, 4 means Marked erythema & Disease is widespread in extent.
Percentage of subjects whose Investigator Global Assessment (IGA) score is decreased by 2 points or more | Weeks 12, 16, 20 and 24
  This assessment is the overall investigator's overall global assessment for the whole body. Minimum 0 to Maximum 4. 0 means No inflammatory signs of atopic dermatitis, 4 means Marked erythema & Disease is widespread in extent.
Score change from Baseline on Pruritus Numerical Rating Scale (NRS) | Weeks 4, 8, 12, 16, 20 and 24
  The NRS is comprised of two items and represents the numbers 0 ("no itch") to 10 ("worst imaginable itch") in the average score of itch and the worst score of itch.
Percentage of subjects whose Pruritus Numerical Rating Scale (NRS) is improved by 3 points or more | Weeks 12, 16, 20 and 24
  The NRS is comprised of two items and represents the numbers 0 ("no itch") to 10 ("worst imaginable itch") in the average score of itch and the worst score of itch.
Percentage change from Baseline in Body Surface Area (BSA) affected by Atopic Dermatitis (AD) | Weeks 4, 8, 12, 16, 20 and 24
  BSA involvement of AD will be assessed for each part of the body using "Wallace rule of nines". This BSA is not calculated by weight and height unlike usual BSA calculation, the Wallace rule of nines is a tool used in pre-hospital and emergency medicine to estimate the total body surface area (BSA) affected by a burn. However, this study, the rule of nines will be used to measure the estimated BSA of atopic dermatitis.
Score change from Baseline in the SCORing Atopic Dermatitis (SCORAD) index | Weeks 4, 8, 12, 16, 20 and 24
  SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). Dermatologists may use this tool before and after treatment to determine whether the treatment has been effective. Maximum value is up to 103 which is the worst outcome.
Score change from Baseline in the Dermatology Life Quality Index (DLQI) | Weeks 4, 8, 12, 16, 20 and 24
  The Dermatology Life Quality Index questionnaire is designed for use in adults. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Score change from Baseline the Patient-Oriented Eczema Measure (POEM) | Weeks 4, 8, 12, 16, 20 and 24
  POEM scores are 0-2 (clear/almost clear); 3-7 (mild); 8-16 (moderate); 17-24 (severe); 25-28 (very severe)
Change from Baseline in biomarker (Immunoglobulin E [IgE]) | Week 4, Week 6, Week 8, Week 12, Week 16, Week 20 and Week 24
  biomarkers will be evaluated from the baseline to each time point. Unit of Measure is IU/mL.
Change from Baseline in biomarker (eosinophil count) | Week 4, Week 6, Week 8, Week 12, Week 16, Week 20 and Week 24
  biomarkers will be evaluated from the baseline to each time point. Unit of measure is cells/μL.
Change from Baseline in biomarker (interleukin [IL]-13) | Week 4, Week 6, Week 8, Week 12, Week 16, Week 20 and Week 24
  biomarkers will be evaluated from the baseline to each time point. Unit of measure is pg/mL.
Change from Baseline in biomarker (interleukin [IL]-17) | Week 4, Week 6, Week 8, Week 12, Week 16, Week 20 and Week 24
  biomarkers will be evaluated from the baseline to each time point. Unit of measure is pg/mL.
Change from Baseline in biomarker (thymus and activation-regulated chemokine [TARC]) | Week 4, Week 6, Week 8, Week 12, Week 16, Week 20 and Week 24
  biomarkers will be evaluated from the baseline to each time point. Unit of measure is pg/mL.
Change from Baseline in biomarker (interleukin [IL]-22) | Week 4, Week 6, Week 8, Week 12, Week 16, Week 20 and Week 24
  biomarkers will be evaluated from the baseline to each time point. Unit of measure is pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Gwang Seong Choi, MD-Ph.D, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No